CLINICAL TRIAL: NCT00115037
Title: Non-Response to Naltrexone (NTX): Next Steps in Managing Alcoholism
Brief Title: Managing Alcoholism in People Who Do Not Respond to Naltrexone
Acronym: EXTEND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, David Oslin, Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAAOSL014851, 708534
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Alcoholism
Keywords: Alcoholism; alcohol abuse; therapy; drug resistance; naltrexone; patient care management; human subject
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Medication Therapy Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase 1 Liberal Response (Experimental): From the start of baseline subjects were randomly assigned to this arm which defined relapse/non-responder as having 5 or heavy drinking days in the first 8 weeks of treatment otherwise the subject was considered a responder.
  Interventions: Drug: Naltrexone
- Phase 1 Stringent Response (Experimental): From the start of baseline subjects were randomly assigned to this arm which defined relapse/non-responder as having 2 or heavy drinking days in the first 8 weeks of treatment otherwise the subject was considered a responder.
  Interventions: Drug: Naltrexone
- Phase 2 nalt and tele for responders (Experimental): Phase 2: Naltrexone and telephone counseling for responders.
  Interventions: Drug: Naltrexone; Behavioral: Telephone Counseling
- Phase 2 nalt, MM and CBI for NR (Experimental): Phase 2: naltrexone, Medication Management (MM) and Combined Behavioral Intervention (CBI) for non-responders (NR).
  Interventions: Drug: Naltrexone; Behavioral: Medication Management (MM); Behavioral: Combined Behavioral Intervention (CBI)
- Phase 2 placebo, MM and CBI for NR (Placebo Comparator): Phase 2: placebo, Medication Management (MM) and Combined Behavioral Intervention (CBI) for non-responders (NR)
  Interventions: Drug: placebo; Behavioral: Medication Management (MM); Behavioral: Combined Behavioral Intervention (CBI)
- Phase 2 naltrexone for responders (Experimental): Phase 2: Naltrexone and TAU for phase 1 responders.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — 100mg/day, up to 8 weeks during Phase 1, 16 weeks in phase 2.
  Other Names: ReVia
  Arms: Phase 1 Liberal Response; Phase 1 Stringent Response; Phase 2 nalt and tele for responders; Phase 2 nalt, MM and CBI for NR; Phase 2 naltrexone for responders
Drug: placebo — placebo comparer for 16 weeks in phase 2.
  Other Names: placebo pill
  Arms: Phase 2 placebo, MM and CBI for NR
Behavioral: Medication Management (MM) — Brief manual-based therapy for up to 8 weeks during phase 1, 16 during phase 2.
  Other Names: MM
  Arms: Phase 2 nalt, MM and CBI for NR; Phase 2 placebo, MM and CBI for NR
Behavioral: Combined Behavioral Intervention (CBI) — 45-60 minute sessions with a certified therapist focused on resolving ambivalence and skill building. Number of sessions guided by achievement of goals identified within treatment plan; minimum 9, maximum 20 sessions over 16 weeks.
  Other Names: CBI
  Arms: Phase 2 nalt, MM and CBI for NR; Phase 2 placebo, MM and CBI for NR
Behavioral: Telephone Counseling — Bi-weekly telephone calls lasting 15-20 minutes focused on the same content as MM.
  Arms: Phase 2 nalt and tele for responders

SUMMARY:
This is a study involving treatment for alcohol dependence (alcoholism). The study will combine motivational enhancement therapy and cognitive behavioral therapy (combined behavioral intervention, or CBI) and tests the benefits of continued/discontinued treatment with naltrexone in a randomized placebo-controlled trial. CBI may have advantages in motivating patients to greater medication adherence and may address psychosocial factors that may limit the effects of naltrexone.

DETAILED DESCRIPTION:
Naltrexone has been established as an efficacious medication to treat alcohol dependence but studies thus far have focused mostly on the acute phase of treatment rather than long-term management and have not offered alternative treatment strategies when patients do not respond to an initial course of naltrexone. For these initial non-responders to naltrexone, it is unclear what adjustments to treatment should be made to increase the likelihood of treatment success. We are unaware of previous research focused specifically on naltrexone non-response. Pilot data from ongoing trials at our center, however, suggest that up to a third of patients fail to respond to naltrexone. Moreover, these non-responsive patients go on to have the worst outcomes during the next 6 months of treatment if maintained on the same combination of naltrexone and medication management (MM). We propose to augment medication management with a combination of motivational enhancement therapy and cognitive behavioral therapy (combined behavioral intervention - CBI) and to test the benefits of continued/discontinued treatment with naltrexone in a randomized placebo-controlled trial. Clinical strategies for second line treatments often favor switching treatments rather than augmentation. However, there may be synergies between naltrexone and CBI that were not apparent with medication management. Specifically, CBI may have advantages in motivating patients to greater medication adherence (a leading cause of naltrexone treatment failure) and CBI may address psychosocial factors that limited or attenuated the effects of naltrexone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current DSM-IV diagnosis of alcohol dependence using the MINI.
* Meets the following drinking criteria as measured by the Timeline Followback (TLFB): * drank within 30 days of randomization; * reports a minimum of 48 standard alcoholic drinks (avg. 12 drinks/wk.) in a consecutive 30-day period over the 90-day period prior to intake; and * has 2 or more days of heavy drinking (defined as over 5 drinks per day in males and over 4 drinks per day in females) in this same pre-treatment period, prior to intake.
* Prior to starting NTX, scores below 8 on the Clinical Inventory of Withdrawal from Alcohol (CIWA), and at least 3 consecutive days of abstinence (2 days abstinence will be permitted with approval by the principal investigator) directly prior to randomization, as determined by Subject report and breathalyzer measures
* Speaks, understands and prints in English.

Exclusion Criteria:

* Has abused or been dependent on opiates in the past 12 months, or evidence of opiate use in month prior to treatment, as assessed by subject report and intake urine drug screen. Use of prescription opioids prior to treatment entry is allowed at the discretion of the investigator. However, subjects must be free from use at the time of randomization.
* Meets DSM IV criteria for current dependence, abuse, or dependence in partial remission on any substance other than alcohol (except nicotine and marijuana). Subjects who test positive on the urine drug screen (with the exception of THC) at the initial visit (a repeat UDSis permitted in cases that are not clear. The repeat UDS should be at least 5 days after the initial test)
* Has a lifetime DSM-IV diagnosis of schizophrenia or any psychotic disorder. Has a current DSM-IV diagnosis of post-traumatic stress disorder (PTST) or bipolar disorder, or any disorder that may interfere with study participation, at the discretion of the investigator.
* Hepatocellular disease indicated by elevations of SGPT (ALT) and SGOT (AST) of at least 5 times normal, or elevated bilirubin (of 1.3 or higher), as evidenced by the most recent lab results prior to randomization. (documentation of Gilberts syndrome will not constitute an exclusion despite elevated bilirubin).
* Has evidence of significant hematological, pulmonary, endocrine, cardiovascular, renal or gastrointestinal disease that the principal investigator considers a risk to participation.
* Has taken any psychotropic medications (or disulfiram) regularly within the last seven days prior to randomization or needs immediate treatment with a psychotropic medication (with the exception of detoxification medications or benadryl used sparingly for sleep). The required washout period for fluoxetine (Prozac®) is 14 days prior to randomization, and the required washout period for other psychotropic medications is 7 days prior to randomization.
* Has taken any detoxification medication on the day of randomization.
* Tests positive on a pregnancy test, is contemplating pregnancy in the next 12 months, is nursing, or is not using an effective contraceptive method if the subject is of child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2003-09; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Treatment Research Center, Chestnut Street, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chakravorty S, Kuna ST, Zaharakis N, O'Brien CP, Kampman KM, Oslin D. Covariates of craving in actively drinking alcoholics. Am J Addict. 2010 Sep-Oct;19(5):450-7. doi: 10.1111/j.1521-0391.2010.00067.x. PMID 20716308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited through advertisements in the local media, referrals from physicians, or self referrals.
Pre-assignment Details: All participants were offered medically monitored outpatient detox as needed.
Groups:
- Phase1: Liberal: Relapse/non-responder defined as having 5 or more heavy drinking days in the first 8 weeks of treatment otherwise the subject was considered a responder.
  Naltrexone: 100mg/day, up to 8 weeks during Phase 1, 16 weeks in phase 2.
- Phase1: Stringent: Relapse/non-responder defined as having 2 or more heavy drinking days in the first 8 weeks of treatment otherwise the subject was considered a responder.
  Naltrexone: 100mg/day, up to 8 weeks during Phase 1, 16 weeks in phase 2.
- Phase2: Responder - Naltx (Usual Care): Phase 2: Naltrexone and TAU for phase 1 responders. Naltrexone: 100mg/day, up to 8 weeks during Phase 1, 16 weeks in phase 2.
- Phase2: Responder - Naltx+Phone (TDM): Phase 2: Naltrexone and telephone counseling for responders. Naltrexone: 100mg/day, up to 8 weeks during Phase 1, 16 weeks in phase 2. Telephone Counseling: Bi-weekly telephone calls lasting 15-20 minutes focused on the same content as MM.
- Phase2: Non-responder - Naltx, MM and CBI: Phase 2: naltrexone, Medication Management (MM) and Combined Behavioral Intervention (CBI) for non-responders (NR).
  Naltrexone: 100mg/day, up to 8 weeks during Phase 1, 16 weeks in phase 2. Medication Management (MM): Brief manual-based therapy for up to 8 weeks during phase 1, 16 during phase 2.
  Combined Behavioral Intervention (CBI): 45-60 minute sessions with a certified therapist focused on resolving ambivalence and skill building. Number of sessions guided by achievement of goals identified within treatment plan; minimum 9, maximum 20 sessions over 16 weeks.
- Phase2: Non-responder - Placebo, MM and CBI: Phase 2: placebo, Medication Management (MM) and Combined Behavioral Intervention (CBI) for non-responders (NR) placebo: placebo comparer for 16 weeks in phase 2. Medication Management (MM): Brief manual-based therapy for up to 8 weeks during phase 1, 16 during phase 2.
  Combined Behavioral Intervention (CBI): 45-60 minute sessions with a certified therapist focused on resolving ambivalence and skill building. Number of sessions guided by achievement of goals identified within treatment plan; minimum 9, maximum 20 sessions over 16 weeks.
Period: Phase1
Arm/Group | Phase1: Liberal | Phase1: Stringent | Phase2: Responder - Naltx (Usual Care) | Phase2: Responder - Naltx+Phone (TDM) | Phase2: Non-responder - Naltx, MM and CBI | Phase2: Non-responder - Placebo, MM and CBI
Started | 152 | 150 | 0 | 0 | 0 | 0
Completed | 127 | 123 | 0 | 0 | 0 | 0
Not Completed | 25 | 27 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 16 | 23 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 4 | 0 | 0 | 0 | 0
Period: Phase2
Arm/Group | Phase1: Liberal | Phase1: Stringent | Phase2: Responder - Naltx (Usual Care) | Phase2: Responder - Naltx+Phone (TDM) | Phase2: Non-responder - Naltx, MM and CBI | Phase2: Non-responder - Placebo, MM and CBI
Started | 0 | 0 | 91 | 92 | 34 | 33
Completed | 0 | 0 | 76 | 77 | 28 | 21
Not Completed | 0 | 0 | 15 | 15 | 6 | 12
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 12 | 14 | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Phase1: Liberal: Definition B of heavy drinker: 5+ days of binge drinking
- Phase1: Stringent: Definition A of heavy drinker: 2+ days of binge drinking
- Total: Total of all reporting groups
Arm/Group | Phase1: Liberal | Phase1: Stringent | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 48.70 (10.40) | 48.49 (10.36) | 48.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 130 | 130 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 146 | 146 | 292
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 45 | 85
  White | 111 | 103 | 214
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Count of Responders and Non-responders in Phase 1
Description: This is the number of patients who responded to phase 1 treatment based on the definition that subjects were randomly assigned to.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Liberal Response: From the start of baseline subjects were randomly assigned to this arm which defined relapse/non-responder as having 5 or more heavy drinking days in the first 8 weeks of treatment otherwise the subject was considered a responder.
  Naltrexone: 100mg/day, up to 8 weeks during Phase 1, 16 weeks in phase 2.
- Phase 1 Stringent Response: From the start of baseline subjects were randomly assigned to this arm which defined relapse/non-responder as having 2 or more heavy drinking days in the first 8 weeks of treatment otherwise the subject was considered a responder.
  Naltrexone: 100mg/day, up to 8 weeks during Phase 1, 16 weeks in phase 2.
Arm/Group | Phase 1 Liberal Response | Phase 1 Stringent Response
Number analyzed (Participants) | 127 | 123
Participants | 103 | 80

2. Primary Outcome: Percentage of Heavy Drinking Days
Description: Percentage of days with heavy drinking, where heavy drinking is 4 (5) or more drinks for females (males) in a 24 hour period.
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: percentage days of heavy drinking
Arm/Group | Phase 2 Naltrexone for Responders | Phase 2 Nalt and Tele for Responders | Phase 2 Nalt, MM and CBI for NR | Phase 2 Placebo, MM and CBI for NR
Number analyzed (Participants) | 83 | 84 | 30 | 27
percentage days of heavy drinking | 0 [0 to 4.8] | 0 [0 to 3.2] | 27.7 [2.8 to 61.6] | 17.8 [0 to 58.7]

ADVERSE EVENTS:
Groups:
- Phase2: Non-responder - Placebo, MM and CBI: Phase 2: placebo, Medication Management (MM) and Combined Behavioral Intervention (CBI) for non-responders (NR) placebo: placebo comparer for 16 weeks in phase 2. Medication Management (MM): Brief manual-based therapy for up to 8 weeks during phase 1, 16 during phase 2.
  Combined Behavioral Intervention (CBI): 45-60 minute sessions with a certified therapist focused on resolving ambivalence and skill building. Number of sessions guided by achievement of goals identified within treatment plan; minimum 9, maximum 20 sessions over 16 wee
Arm/Group | Phase1: Liberal | Phase1: Stringent | Phase2: Responder - Naltx (Usual Care) | Phase2: Responder - Naltx+Phone (TDM) | Phase2: Non-responder - Naltx, MM and CBI | Phase2: Non-responder - Placebo, MM and CBI
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/150 | 1/91 | 0/92 | 0/34 | 1/33
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/150 | 0/91 | 0/92 | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/152 | 0/150 | 0/91 | 0/92 | 0/34 | 0/33

LIMITATIONS AND CAVEATS:
Overall the sample size was limited for detecting results in the second phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No